CLINICAL TRIAL: NCT03946254
Title: Effect of Strength Training on Executive Functions in Elderly People With Mild Cognitive Impairment
Acronym: Executive-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Manuel Jesús, Science of physical activity and sport, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: University of seville
Record Dates: First submitted 2019-05-03; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Strength Training; Executive Function

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: After the random assignment of the groups, the coaches will be oblivious to the investigation, so there is no bias.Furthermore, the principal investigator will not know where the data of each group comes from.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): THE EXPERIMENTAL GROUP WILL DEVELOP 20 WEEKS OF TRAINING TO IMPROVE THE MUSCLE CAPACITY. FOR THIS, FORCE EXERCISES WILL BE DEVELOPED IN GUIDED MACHINES.
  Interventions: Other: Effect of strength training on executive functions in elderly people with mild cognitive impairment.
- Control (Experimental): THE CONTROL GROUP WILL DEVELOP 20 WEEKS OF BALANCE AND BREATHING EXERCISES.
  Interventions: Other: Effect of strength training on executive functions in elderly people with mild cognitive impairment.

INTERVENTIONS:
Other: Effect of strength training on executive functions in elderly people with mild cognitive impairment. — Strength training sessions will have a frequency of 3 times per week (Monday, Tuesday and Wednesday) for 20 weeks. In addition, each subject is subject to an individualized training program according to the workload in order to progressively increase the intensity of work. The workload will be modified progressively by influencing both the total volume of repetitions and the intensity of the exercises. The exercises will be controlled movements and not harmful, as guided machines will be used to facilitate the execution of actions. In addition, the largest amount of muscle groups to be able to generate strength gains in all muscle groups. The control group will perform breathing exercises and low intensity stretching during the same days and with the same duration as the experimental group

SUMMARY:
Cognitive impairment or dementia is their last degree in one of the main concerns at a social level in these ages. To this day, there are different pharmacological and non-pharmacological therapies that can help prevent deterioration, as in this case, physical exercise.

In the existing scientific literature, you can find a lot of information about the effect of aerobic exercise on cognition, but little is known about the effect of force exercise and its effect on general cognition and executive functions.

Therefore, in this research the investigators will investigate the effect of strength training in people over 60 with a diagnosis of mild cognitive impairment in executive functions. For this, a controlled and randomized clinical trial will be developed in the city of Seville

DETAILED DESCRIPTION:
The training program will last 20 weeks and a frequency of 3 times / week.

During the week 0 the initial evaluation will be developed. Between weeks 1-20, the training program will be addressed. In week 21, all the changes made in all the measured variables will be evaluated.

Finally, in week 33 the variables will be measured again to see if the possible improvements given in the training program last over time.

The experimental group will perform a planned and individualized training with guided machines and training loads will be adjusted at the beginning of each week.

The control group will perform breathing and relaxation exercises to avoid a sample death.

After the intervention, there will be a follow-up phase for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* The sample is made up of people over 60 years of age, who are not active professionally, speak and understand the Spanish language.
* In addition, they should be diagnosed with mild cognitive impairment. This will be evaluated by specialists through the minimental test (score between 24 and 28).
* On the other hand, they should not suffer from other serious psychiatric or neurodegenerative neurological diseases.
* In relation to mental health, it will be a reason for exclusion to have had 3 episodes of depression in the last 5 years or 10 episodes that have required some psychiatric or medical treatment.In addition,
* The people included must be postmenopausal

Exclusion Criteria:

* Participate in other physical exercise programs in a systematic way or in individualized and systematic programs in cognitive programs.
* Dispose of cardiovascular diseases, heart diseases that involve an absolute contradiction of physical exercise (unstable angina, severe auroventricular block) and cerebrovascular or have suffered a heart attack in the last 6 years.
* Have had seizures (More than 2 in the last 12 months).
* Consumption of alcohol 20 grams / day or 2 beers or wine glasses daily.
* Functional limitations (According to Functional activities Questionnaire)
* Being a musician or bilingual.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Baseline of Inhibitory control | week 0
  To measure the inhibitory control, the "Stroop test" will be used. It is a short test and consists of 3 parts. In the first part they must read the greatest number of words in a sheet with a total of 100 words that appear in 5 columns. For 45 seconds they should read the largest number of words. At the end of the time the number will be written down of words read. Next, they should identify colors from a list of symbols without meaning, but colored in different colors. The subject will have to identify and name the greatest number of colors.
  Finally, the subject is given a list of words with the name of colors, but written with a different color from the one the word refers to.This test aims to assess the inhibitory control.
Mean Change from Baseline in Inhibitory control | week 21
  To measure the inhibitory control, the "Stroop test" will be used. It is a short test and consists of 3 parts. In the first part they must read the greatest number of words in a sheet with a total of 100 words that appear in 5 columns. For 45 seconds they should read the largest number of words. At the end of the time the number will be written down of words read. Next, they should identify colors from a list of symbols without meaning, but colored in different colors. The subject will have to identify and name the greatest number of colors.
  Finally, the subject is given a list of words with the name of colors, but written with a different color from the one the word refers to.This test aims to assess the inhibitory controlof words read.
Inhibitory control in the follow-up phase | week 33
  To measure the inhibitory control, the "Stroop test" will be used. It is a short test and consists of 3 parts. In the first part they must read the greatest number of words in a sheet with a total of 100 words that appear in 5 columns. For 45 seconds they should read the largest number of words. At the end of the time the number will be written down of words read. Next, they should identify colors from a list of symbols without meaning, but colored in different colors. The subject will have to identify and name the greatest number of colors.
  Finally, the subject is given a list of words with the name of colors, but written with a different color from the one the word refers to.This test aims to assess the inhibitory controlof words read.

SECONDARY OUTCOMES:
Baseline of general cognition | Week 0
  Global cognition is evaluated through the mini-mental test (Folstein, Folstein, & McHugh, 1975). It is a brief and quick test to apply and is frequently used to diagnose the degree of cognitive decline. It should be noted how various variables such as the socio-educational level, and age among others, can affect the result. In addition, the mini-mental test is low cost and can be applied by any professional with a minimum of knowledge and training towards their development. The diagnostic values for mild cognitive impairment are between 24 and 28.
Mean Change from Baseline in General cognition | week 21
  Global cognition is evaluated through the mini-mental test (Folstein, Folstein, & McHugh, 1975). It is a brief and quick test to apply and is frequently used to diagnose the degree of cognitive decline. It should be noted how various variables such as the socio-educational level, and age among others, can affect the result. In addition, the mini-mental test is low cost and can be applied by any professional with a minimum of knowledge and training towards their development. The diagnostic values for mild cognitive impairment are between 24 and 28.
General cognition in the follow-up phase | week 33
  Global cognition is evaluated through the mini-mental test (Folstein, Folstein, & McHugh, 1975). It is a brief and quick test to apply and is frequently used to diagnose the degree of cognitive decline. It should be noted how various variables such as the socio-educational level, and age among others, can affect the result. In addition, the mini-mental test is low cost and can be applied by any professional with a minimum of knowledge and training towards their development. The diagnostic values for mild cognitive impairment are between 24 and 28.
Baseline of physical condition | week 0
  Senior Fitness Test. This test battery allows us to evaluate the physical condition of elderly people safely. This battery can develop in ages from 60 to 94 years, encompassing various levels of physical and functional capacity (Rikli & Jones, 1999).Due to its easy application, no specific material is required for its development, so it can be developed outside the laboratory.
  This test battery consists of 7 tests: The tests described here are quantified by the distance achieved.
  Test of flexibility of the lower extremities, Put your hands behind your back, Get up and walk and sit down again.
  In all the tests, the distance or number of repetitions made will be noted to later make comparisons with reference tables already established according to the ages.
Mean Change from Baseline in Physical condition | week 21
  Senior Fitness Test. This test battery allows us to evaluate the physical condition of elderly people safely. This battery can develop in ages from 60 to 94 years, encompassing various levels of physical and functional capacity (Rikli & Jones, 1999).Due to its easy application, no specific material is required for its development, so it can be developed outside the laboratory.
  This test battery consists of 7 tests: The tests described here are quantified by the distance achieved.
  Test of flexibility of the lower extremities, Put your hands behind your back, Get up and walk and sit down again.
  In all the tests, the distance or number of repetitions made will be noted to later make comparisons with reference tables already established according to the ages.
Physical condition in the follow-up phase | week 33
  Senior Fitness Test. This test battery allows us to evaluate the physical condition of elderly people safely. This battery can develop in ages from 60 to 94 years, encompassing various levels of physical and functional capacity (Rikli & Jones, 1999).Due to its easy application, no specific material is required for its development, so it can be developed outside the laboratory.
  This test battery consists of 7 tests: The tests described here are quantified by the distance achieved.
  Test of flexibility of the lower extremities, Put your hands behind your back, Get up and walk and sit down again.
  In all the tests, the distance or number of repetitions made will be noted to later make comparisons with reference tables already established according to the ages.
Baseline of physical condition variante | week 0
  Senior Fitness Test. This test battery allows us to evaluate the physical condition of elderly people safely. This battery can develop in ages from 60 to 94 years, encompassing various levels of physical and functional capacity (Rikli & Jones, 1999).Due to its easy application, no specific material is required for its development, so it can be developed outside the laboratory.
  This test battery consists of 7 tests. The tests described here are quantified by the maximum number of repetitions performed.
  Sit and get up from a chair for 30 seconds, push-ups for 30 seconds, In all the tests, the distance or number of repetitions made will be noted to later make comparisons with reference tables already established according to the ages.
Mean Change from Baseline in Physical condition variante | week 21
  Senior Fitness Test. This test battery allows us to evaluate the physical condition of elderly people safely. This battery can develop in ages from 60 to 94 years, encompassing various levels of physical and functional capacity (Rikli & Jones, 1999).Due to its easy application, no specific material is required for its development, so it can be developed outside the laboratory.
  This test battery consists of 7 tests. The tests described here are quantified by the maximum number of repetitions performed.
  Sit and get up from a chair for 30 seconds, push-ups for 30 seconds, In all the tests, the distance or number of repetitions made will be noted to later make comparisons with reference tables already established according to the ages.
Physical condition variante in the follow-up phase | week 33
  Senior Fitness Test. This test battery allows us to evaluate the physical condition of elderly people safely. This battery can develop in ages from 60 to 94 years, encompassing various levels of physical and functional capacity (Rikli & Jones, 1999).Due to its easy application, no specific material is required for its development, so it can be developed outside the laboratory.
  This test battery consists of 7 tests. The tests described here are quantified by the maximum number of repetitions performed.
  Sit and get up from a chair for 30 seconds, push-ups for 30 seconds, In all the tests, the distance or number of repetitions made will be noted to later make comparisons with reference tables already established according to the ages.
Baseline of blood test | week 0
  Only 15 ml of blood will be extracted from the antecubital vein to measure the concentrations of different biochemical parameters, such as the BDFN and IGF-1. To avoid interferences in the blood analysis, it is necessary that the patient goes on an empty stomach. It is also necessary that during the previous day the participant fulfills a normal sleep monitoring cycle and that he does not eat chocolate, cocoa, tea, coffee or any other stimulant.
Mean Change from Baseline in Blood test | week 21
  Only 15 ml of blood will be extracted from the antecubital vein to measure the concentrations of different biochemical parameters, such as the BDFN and IGF-1. To avoid interferences in the blood analysis, it is necessary that the patient goes on an empty stomach. It is also necessary that during the previous day the participant fulfills a normal sleep monitoring cycle and that he does not eat chocolate, cocoa, tea, coffee or any other stimulant.
Baseline of strength | week 0
  The point of maximum power is an elaborate and accurate assessment of muscle strength and is often evaluated at a speed of 60º per second. Therefore, the Biodex 4 system will be used to assess the capacity to generate the power peak of each subjectby knee extension.
Mean Change from Baseline in Strength | week 21
  The point of maximum power is an elaborate and accurate assessment of muscle strength and is often evaluated at a speed of 60º per second. Therefore, the Biodex 4 system will be used to assess the capacity to generate the power peak of each subjectby knee extension.
Strength in the follow-up phase | week 33
  The point of maximum power is an elaborate and accurate assessment of muscle strength and is often evaluated at a speed of 60º per second. Therefore, the Biodex 4 system will be used to assess the capacity to generate the power peak of each subjectby knee extension.
Baseline of cognitive flexibility | week 0
  To evaluate the cognitive flexibility, will be used the WISCONSIN TEST. This test consists of two sets of 64 cards. The letters present various combinations according to 4 geometric shapes, 4 colors and 4 quantities.
Mean Change from Baseline in cognitive flexibility | week 21
  To evaluate the cognitive flexibility, will be used the WISCONSIN TEST. This test consists of two sets of 64 cards. The letters present various combinations according to 4 geometric shapes, 4 colors and 4 quantities.
cognitive flexibility in the follow-up phase | week 33
  To evaluate the cognitive flexibility, will be used the WISCONSIN TEST. This test consists of two sets of 64 cards. The letters present various combinations according to 4 geometric shapes, 4 colors and 4 quantities.
Baseline of cognitive flexibility variante | week 0
  "Trail Making test part B" will be used to assess cognitive flexibility. This reliable test and valid consists of a page where you must surround numbers and letters. The numbers are they extend from 1 to 13 and the letters from A to L.
Mean Change from Baseline in cognitive flexibility variante | week 21
  "Trail Making test part B" will be used to assess cognitive flexibility. This reliable test and valid consists of a page where you must surround numbers and letters. The numbers are they extend from 1 to 13 and the letters from A to L.
cognitive flexibility variante in the follow-up phase | week 33
  "Trail Making test part B" will be used to assess cognitive flexibility. This reliable test and valid consists of a page where you must surround numbers and letters. The numbers are they extend from 1 to 13 and the letters from A to L.
Baseline of working memory | week 0
  For that, wi will used the Verbal digit span forward and backward tests.This test is an excellent tool to evaluate working memory. The examiner reads a sequence of numbers and the participant must repeat it. It is composed of two parts, direct or indirect. In the first the subject must say the sequence of numbers in the order they appear. On the other hand, the indirect must name the numbers that appeared in reverse order. The length of the sequences of numbers increases progressively and two sequences with the same number are always administered. The task is suspended when the subject fails twice in the same sequence. This test gives us a measure of the attention capacity and working memory.
Mean Change from Baseline in working memory | week 21
  For that, wi will used the Verbal digit span forward and backward tests.This test is an excellent tool to evaluate working memory. The examiner reads a sequence of numbers and the participant must repeat it. It is composed of two parts, direct or indirect. In the first the subject must say the sequence of numbers in the order they appear. On the other hand, the indirect must name the numbers that appeared in reverse order. The length of the sequences of numbers increases progressively and two sequences with the same number are always administered. The task is suspended when the subject fails twice in the same sequence. This test gives us a measure of the attention capacity and working memory.
Working memory in the follow-up phase | week 33
  For that, wi will used the Verbal digit span forward and backward tests.This test is an excellent tool to evaluate working memory. The examiner reads a sequence of numbers and the participant must repeat it. It is composed of two parts, direct or indirect. In the first the subject must say the sequence of numbers in the order they appear. On the other hand, the indirect must name the numbers that appeared in reverse order. The length of the sequences of numbers increases progressively and two sequences with the same number are always administered. The task is suspended when the subject fails twice in the same sequence. This test gives us a measure of the attention capacity and working memory.

CONTACTS AND LOCATIONS:
Overall Officials: manuel jesus j roldan, Sports Sci, Principal Investigator — University of Seville
Locations (1):
- Education Faculty, Seville, Spain

IPD SHARING:
Plan to Share IPD: No